CLINICAL TRIAL: NCT00931255
Title: Delayed Tacrolimus to Sirolimus Conversion in Renal Transplant Recipients With Delayed Graft Function
Brief Title: Tacrolimus to Sirolimus Conversion for Delayed Graft Function
Acronym: RAPA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was stopped because of slow recruitment.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Abdoleza Haririan, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00042201
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Kidney Transplant; Delayed Graft Function
Keywords: kidney transplant; tacrolimus; sirolimus; delayed graft function; Graft survival; Acute rejection; Chronic allograft nephropathy
MeSH Terms: conditions — Delayed Graft Function | interventions — Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): Tacrolimus will be continued with target 12-hour trough level 7-10 ng/ml (tandem mass spectrometry) during the first year and 5-8 during second year.
  Interventions: Drug: Tacrolimus
- Sirolimus (Active Comparator): 5 mg, PO , daily
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Tacrolimus — 3-10 mg, PO, BID based on 12 hour trough on serum blood levels, adjusted according to protocol
  Other Names: FK506, Prograf
  Arms: Tacrolimus
Drug: Sirolimus — 5 mg, PO, daily based on 24 hour serum blood levels, adjusted according to protocol
  Other Names: Rapamune, Rapamycin
  Arms: Sirolimus

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of conversion from tacrolimus to sirolimus early after kidney transplantation in patients with delayed graft function (DGF)and slow graft function (SGF) in improving graft function and delaying chronic allograft nephropathy. The investigators hypothesize that conversion from tacrolimus to sirolimus in renal transplant recipients with DGF/SGF in early months after surgery will improve graft function and decrease the progression of graft fibrosis.

DETAILED DESCRIPTION:
Eligible study subjects will be randomized into two groups 8-18 weeks after surgery. One group will be maintained on tacrolimus according to the standard of care at our center. In the second group tacrolimus will be converted to sirolimus, with one week overlap between sirolimus therapy and tacrolimus taper. All the deceased donor kidney transplant recipients transplanted at our center who experience DGF/SGF are eligible for inclusion in this study, if they meet the inclusion/exclusion criteria as detailed later.

Data will be collected on patient demographics, duration on dialysis, history of diabetes and chronic hepatitis C, previous transplantation, PRA, donor source, warm and cold ischemia time, donor demographics and comorbidity such as diabetes and hypertension, serum creatinine at the time of organ removal, early graft function, number of dialysis treatments after transplantation, induction agent and immunosuppressive regimen including the dose or level of the drugs at 3, 6, 9, 12, 18, and 24 months. Similar data regarding use of ACE inhibitors/ARBs, erythropoietic agents, number of anti-hypertensives and lipid lowering agents will be collected. In addition, the following tests and procedures will be obtained for this study.

1. GFR measurement by cold iothalamate method at one year after transplantation.
2. Evaluation of routine surveillance graft biopsies for chronic changes at 3 and 12 months posttransplant by morphometric analysis.
3. Spot urine protein, albumin, and creatinine measurement at 3 and 12 months.
4. Estimate GFR at 3, and 12 months using MDRD, CG, and Nankivell formulas
5. Examine the surveillance and indicated biopsies for acute rejection and BK nephropathy.
6. Fasting lipid profile at 3 and 12 months for all patients, and 24 months for those with at least 2 years of follow up.
7. Office blood pressure measurements at 3 and 12 months for all patients, and 24 months for those with at least 2 years of follow up.
8. Measurement of CRP, IL-6, and MCP at 3 and 12 months.

The safety measures will include:

Incidence of leukopenia (WBC < 3000) or thrombocytopenia (PLT < 100,000); hemoglobin level at 12 months; proteinuria at 12 months; incidence of oral aphthous ulcers; incidence of new onset diabetes, incidence of CMV infection and rate of drug withdrawal due to side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age => 18.
2. Recipient of a deceased donor kidney transplant.
3. Delayed graft function, defined as need for dialysis during first week after surgery or slow graft function, defined as creatinine >=3.0 by post-op day 5 without requiring dialysis
4. Stable serum creatinine for 2 weeks prior to enrollment.
5. Able to give informed consent.
6. Compliant with medical regimen and clinic visits.

Exclusion Criteria:

1. Episode of acute rejection within 4 weeks prior to enrollment.
2. Calculated GFR < 30 ml/min.
3. Interstitial fibrosis & tubular atrophy in transplant biopsy higher than grade II (Banff"05 update).
4. Proteinuria > 500 mg/24 h or spot urine protein/creatinine > 0.5.
5. Total fasting cholesterol level > 300 mg/dl or triglyceride > 500 mg/dl despite optimal lipid lowering therapy.
6. Recipient of pancreas or liver allografts.
7. Leukopenia (WBC < 3000 mm3) within 2 weeks prior to enrollment.
8. Leukopenia (WBC < 2000 mm3) within 4 weeks prior to enrollment.
9. Thrombocytopenia (platelets count < 100,000/mm3) within 2 weeks prior to enrollment.
10. Unwilling to comply with study protocol.
11. Enrollment in another drug trial that precludes use of sirolimus.
12. Diagnosis of malignancy within 2 years prior to enrollment, except adequately treated non-melanoma skin cancer.
13. For women, pregnancy.
14. Allergy to iodine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdolreza Haririan, MD, MPH, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus | Sirolimus
Started | 17 | 15
Completed | 15 | 12
Not Completed | 2 | 3
Not completed — Follow up biopsy not done | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Sirolimus | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.7) | 49.9 (10.1) | 51.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Composite Endpoint of Reduction of e eGFR at One Year by More Than 15% & the Progression in Fibrosis Score at One Year by >=20% Compared With the Baseline Values
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 15 | 12
participants | 6 | 9

2. Secondary Outcome: eGFR
Time Frame: One year
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
mL/min per 1.73 m^2 | 56.4 (15.2) | 53.7 (19.2)

3. Secondary Outcome: Change in eGFR From Baseline to 1-year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
mL/min per 1.73 m^2 | 7.45 (11.5) | 1.57 (10.7)

4. Secondary Outcome: Graft Survival (Actual, Actuarial)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
participants | 16 | 14

5. Secondary Outcome: Incidence of Acute Rejection (Actual, Actuarial)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
participants | 1 | 1

6. Secondary Outcome: Incidence of BK Nephropathy (Cumulative)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
participants | 1 | 0

7. Secondary Outcome: Change in Inflammatory Marker : CRP From Baseline
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
mg/L | -1668 (9403) | 4510 (14495)

8. Secondary Outcome: Change in Inflammatory Marker, IL-6 From Baseline
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
pg/mL | -0.7 (8.53) | 6.2 (14.1)

9. Secondary Outcome: Change in Inflammatory Marker, MCP, From Baseline
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus | Sirolimus
Number analyzed (Participants) | 17 | 15
pg/mL | -787.5 (693.9) | -965.2 (753.6)

ADVERSE EVENTS:
Arm/Group | Tacrolimus | Sirolimus
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 1/17 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (N=17) | Sirolimus (N=15)
CMV viremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was stopped because of slow enrollment. Hence, the target enrollment number was not achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No